CLINICAL TRIAL: NCT00894543
Title: Menopause Strategies: Finding Lasting Answers for Symptoms and Health: Efficacy of a Selective Serotonin Reuptake Inhibitor (SSRI) for Menopausal Symptoms in Midlife Women
Brief Title: MsFLASH-01: Escitalopram for Menopausal Symptoms in Midlife Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Andrea LaCroix, Garnet Anderson, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MsFLASH-01; 1U01AG032699-01 (NIH); 1U01AG032656-01 (NIH)
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Hot Flashes; Menopause; Vasomotor Symptoms
Keywords: Hot flashes; Menopause; Vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Active Comparator): Escitalopram is a selective serotonin reuptake inhibitor (SSRI)
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Inactive pill
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Escitalopram — 10 mg (1 pill) escitalopram daily for the first four weeks. Dose increased to 20 mg (2 pills) escitalopram daily if relief from hot flashes has not occurred during the first four weeks of the daily 10 mg dose.
  Other Names: Lexapro®.
  Arms: Escitalopram
Other: Placebo — Inactive pill (1 pill or 2 pills) daily for the 8-11 weeks of the trial.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether a medication reduces the number, severity and bothersomeness of menopausal hot flashes. Escitalopram (also called Lexapro®) is a selective serotonin reuptake inhibitor (SSRI). It is sold by prescription for depression and general anxiety disorder. An SSRI increases serotonin, a brain substance that is believed to influence mood. Serotonin may also affect brain levels of estradiol, a hormone related to hot flashes. This research study will test whether escitalopram reduces menopausal hot flashes.

DETAILED DESCRIPTION:
The MsFLASH-01 study, Efficacy of a Selective Serotonin Reuptake Inhibitor (SSRI) for Menopausal Symptoms in Midlife Women is a randomized, double-blind, placebo-controlled, parallel arm clinical trial. The design includes: 3 weeks of daily recording of hot flashes prior to drug treatment; 8 weeks of double-blind treatment with escitalopram or placebo with dose escalation at 4 weeks among non-responders; 1 week of drug taper for those on higher dose, followed by 2 weeks with no treatment; and a telephone follow-up post-treatment. This study is one of five clinical trials to be conducted as part of the Menopause Strategies - Finding Lasting Answers for Symptoms and Health (MsFLASH) study, a network of investigators and clinical trials designed to find new ways to alleviate the most common, bothersome symptoms of the menopausal transition.

ELIGIBILITY:
Inclusion Criteria, Common to all MsFLASH Studies:

* Females aged 40-62 years.
* Menopausal, including:

  * Women with a uterus who have skipped 2 or more menstrual cycles with an amenorrhea interval ≥60 days in the past 12 months.
  * Women who have had a bi-lateral oophorectomy (surgical removal of both ovaries).
  * Women without a uterus who still have ovaries, under certain conditions determined during screening.
* Having bothersome hot flashes.
* In general good health as determined by medical history and physical measures.
* Signed informed consent.

Exclusion Criteria, Common to all MsFLASH Studies:

* Use of hormone therapy or hormonal contraceptives during the 2 months before enrollment and for the duration of the study. Certain exceptions apply, determined during screening.
* Use of any other therapy that is taken specifically for hot flashes, including prescription, over-the-counter, or herbal therapies in the past month and duration of the study.
* Any current severe or unstable medical illness.
* Uncontrolled hypertension (>160/100) or resting heart rate >110.
* History of endometrial or ovarian cancer; MI, angina, or cerebrovascular events.
* Pregnancy, intending pregnancy, breast feeding.
* Current participation in another drug trial or intervention study.
* Inability or unwillingness to complete the study procedures.
* Certain other conditions, determined during screening.

Exclusion Criteria, Specific to MsFLASH-01:

* Use of selective estrogen receptor modulators (SERMS) or aromatase inhibitors during the two months before enrollment.
* Use of gabapentin, pregabalin, triptans, warfarin (Coumadin®), or St. John's Wort.
* Known hypersensitivity to escitalopram (Lexapro®) or citalopram (Celexa®).
* Use of antidepressants during the past 30 days before starting Study 01, including SSRIs, serotonin-norepinephrine reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MAOIs), and anxiolytics.
* Not using a medically approved method of birth control, if sexually active and not 12 or more months since last menstrual period.
* History of liver, gall bladder, renal disease, or uncontrolled seizure disorder.
* Certain other conditions, determined during screening.

Ages: 40 Years to 62 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W Freeman, PhD, Principal Investigator — University of Pennsylvania Medical Center; Andrea Z LaCroix, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Garnet L Anderson, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Kris Ensrud, MD, Study Chair — University of Minnesota
Locations (5):
- United States (5):
  - Northern California Kaiser, Division of Research, Oakland, California
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Harvard Medical School, Boston, Massachusetts
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Freeman EW, Guthrie KA, Caan B, Sternfeld B, Cohen LS, Joffe H, Carpenter JS, Anderson GL, Larson JC, Ensrud KE, Reed SD, Newton KM, Sherman S, Sammel MD, LaCroix AZ. Efficacy of escitalopram for hot flashes in healthy menopausal women: a randomized controlled trial. JAMA. 2011 Jan 19;305(3):267-74. doi: 10.1001/jama.2010.2016. PMID 21245182
- [Result] Carpenter JS, Guthrie KA, Larson JC, Freeman EW, Joffe H, Reed SD, Ensrud KE, LaCroix AZ. Effect of escitalopram on hot flash interference: a randomized, controlled trial. Fertil Steril. 2012 Jun;97(6):1399-404.e1. doi: 10.1016/j.fertnstert.2012.03.001. Epub 2012 Apr 3. PMID 22480818
- [Result] Ensrud KE, Joffe H, Guthrie KA, Larson JC, Reed SD, Newton KM, Sternfeld B, Lacroix AZ, Landis CA, Woods NF, Freeman EW. Effect of escitalopram on insomnia symptoms and subjective sleep quality in healthy perimenopausal and postmenopausal women with hot flashes: a randomized controlled trial. Menopause. 2012 Aug;19(8):848-55. doi: 10.1097/gme.0b013e3182476099. PMID 22433978
- [Result] Reed SD, Guthrie KA, Joffe H, Shifren JL, Seguin RA, Freeman EW. Sexual function in nondepressed women using escitalopram for vasomotor symptoms: a randomized controlled trial. Obstet Gynecol. 2012 Mar;119(3):527-38. doi: 10.1097/AOG.0b013e3182475fa4. PMID 22353950
- [Result] LaCroix AZ, Freeman EW, Larson J, Carpenter JS, Joffe H, Reed SD, Newton KM, Seguin RA, Sternfeld B, Cohen L, Ensrud KE. Effects of escitalopram on menopause-specific quality of life and pain in healthy menopausal women with hot flashes: a randomized controlled trial. Maturitas. 2012 Dec;73(4):361-8. doi: 10.1016/j.maturitas.2012.09.006. Epub 2012 Sep 30. PMID 23031421
- [Result] Joffe H, Guthrie KA, Larson J, Cohen LS, Carpenter JS, Lacroix AZ, Freeman EW. Relapse of vasomotor symptoms after discontinuation of the selective serotonin reuptake inhibitor escitalopram: results from the menopause strategies: finding lasting answers for symptoms and health research network. Menopause. 2013 Mar;20(3):261-8. doi: 10.1097/GME.0b013e31826d3108. PMID 23435022
- [Derived] Diem SJ, LaCroix AZ, Reed SD, Larson JC, Newton KM, Ensrud KE, Woods NF, Guthrie KA. Effects of pharmacologic and nonpharmacologic interventions on menopause-related quality of life: a pooled analysis of individual participant data from four MsFLASH trials. Menopause. 2020 Oct;27(10):1126-1136. doi: 10.1097/GME.0000000000001597. PMID 32701665
- [Derived] Guthrie KA, Larson JC, Ensrud KE, Anderson GL, Carpenter JS, Freeman EW, Joffe H, LaCroix AZ, Manson JE, Morin CM, Newton KM, Otte J, Reed SD, McCurry SM. Effects of Pharmacologic and Nonpharmacologic Interventions on Insomnia Symptoms and Self-reported Sleep Quality in Women With Hot Flashes: A Pooled Analysis of Individual Participant Data From Four MsFLASH Trials. Sleep. 2018 Jan 1;41(1):zsx190. doi: 10.1093/sleep/zsx190. PMID 29165623
- [Derived] Guthrie KA, LaCroix AZ, Ensrud KE, Joffe H, Newton KM, Reed SD, Caan B, Carpenter JS, Cohen LS, Freeman EW, Larson JC, Manson JE, Rexrode K, Skaar TC, Sternfeld B, Anderson GL. Pooled Analysis of Six Pharmacologic and Nonpharmacologic Interventions for Vasomotor Symptoms. Obstet Gynecol. 2015 Aug;126(2):413-422. doi: 10.1097/AOG.0000000000000927. PMID 26241433
- [Derived] Newton KM, Carpenter JS, Guthrie KA, Anderson GL, Caan B, Cohen LS, Ensrud KE, Freeman EW, Joffe H, Sternfeld B, Reed SD, Sherman S, Sammel MD, Kroenke K, Larson JC, Lacroix AZ. Methods for the design of vasomotor symptom trials: the menopausal strategies: finding lasting answers to symptoms and health network. Menopause. 2014 Jan;21(1):45-58. doi: 10.1097/GME.0b013e31829337a4. PMID 23760428

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from July 2009 to June 2010. The trial was conducted at four MsFLASH network sites: University of Pennsylvania, Massachusetts General Hospital, Indiana University, Kaiser Permanente Division of Research in Oakland, California
Pre-assignment Details: Following enrollment (signing the consent), symptoms and health were reviewed, brief physical exam conducted and urine pregnancy test administered, daily hot flash diaries completed for one week (in addition to two weeks before enrollment).
Groups:
- Escitalopram: Escitalopram is a selective serotonin reuptake inhibitor (SSRI). For the first four weeks, participants took 1 pill daily (escitalopram 10 mg or placebo). At 4 weeks, if hot flash frequency was not reduced by at least 50% or there was no decrease in severity, the dose was increased to 2 pills daily(escitalopram 20 mg or placebo) unless precluded by unacceptable adverse events. At 8 weeks, participants taking 1 pill per day stopped treatment; participants taking 2 pills per day tapered the dose over a week.
Period: Baseline
Arm/Group | Escitalopram | Placebo
Started | 104 | 101
Completed | 104 | 101
Not Completed | 0 | 0
Period: Baseline to Week 4
Arm/Group | Escitalopram | Placebo
Started | 104 | 101
Completed | 101 | 99
Not Completed | 3 | 2
Not completed — No diary or lost or withdrew | 3 | 2
Period: Week 4 to Week 8
Arm/Group | Escitalopram | Placebo
Started | 101 | 99
Completed | 97 | 97
Not Completed | 4 | 2
Not completed — No diary or lost or withdrew | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 104 | 101 | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 104 | 101 | 205
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53.45 (4.20) | 54.36 (3.86) | 53.9 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 101 | 205
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 48 | 95
  White | 53 | 49 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 104 | 101 | 205
Menopausal Status [Number; unit: participants]
  Postmenopause | 84 | 83 | 167
  Late transition | 17 | 15 | 32
  Early transition | 3 | 3 | 6
Body Mass Index (BMI) [Number; unit: participants] — BMI calculated as (body weight in kilograms) divided by (body height in meters squared) (kg/m^2)
  participants
    <25, kg/m^2 | 32 | 22 | 54
    25-<30, kg/m^2 | 34 | 38 | 72
    >=30, kg/m^2 | 38 | 40 | 78
    Missing data | 0 | 1 | 1
Hysterectomy [Number; unit: participants]
  Hysterectomy | 13 | 13 | 26
  Hysterectomy and oophorectomy | 11 | 8 | 19
  Oophorectomy only | 3 | 1 | 4
  None | 77 | 78 | 155
  Don't know | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Daily Frequency of Hot Flashes Per Day Assessed by Prospective Daily Diaries
Description: Baseline hot flash frequency per day was calculated as the daily mean of the daily totals reported during the first two screening weeks.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: Hot flashes/day
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 104 | 101
Hot flashes/day | 9.88 [8.67 to 11.10] | 9.66 [8.70 to 10.63]

2. Secondary Outcome: Daily Hot Flash Bother, Recorded on Daily Diaries
Description: Daily Hot flash bother scores were calculated by selecting the highest bother rating for hot flashes or night sweats for each woman in each 24-hour day. The score was set to missing on on any day data were missing or or hot flashes equaled 0. The daily mean of daily ratings for the first 2 screening weeks is reported.
  Hot flash bother was rated as 1 (none), 2 (a little), 3 (moderately), or 4 (a lot) as adopted from the Study of Women Across the Nation (SWAN).
Time Frame: Baseline
Population: Twice daily rating for bother using response categories from the Study of Women Across the Nation (SWAN): 1 (not at all), 2 (very little), 3 (moderately), 4 (a lot).
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 104 | 101
Scores on a scale | 3.12 [3.03 to 3.22] | 3.16 [3.06 to 3.26]

3. Primary Outcome: Change in Daily Frequency of Hot Flashes Between Baseline and Week 4 as Assessed by Prospective Daily Diaries
Description: Change in daily hot flash frequency was calculated as the daily mean difference between baseline and week 4. Baseline was calculated as the daily mean of the daily frequencies for the first two screening weeks. Week 4 was calculated as the daily mean of the daily frequencies during the week prior to the week 4 visit.
Time Frame: week 4 minus baseline
Measure: Mean (95% Confidence Interval); unit: Hot flashes/day
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 101 | 99
Hot flashes/day | -4.37 [-5.24 to -3.50] | -2.49 [-3.31 to -1.66]

4. Primary Outcome: Change in Daily Frequency of Hot Flashes Between Baseline and Week 8 as Assessed by Prospective Daily Diaries
Description: Change in daily hot flash frequency was calculated as the daily mean difference between baseline and week 8. Baseline was calculated as the daily mean of the frequencies for the first two screening weeks. Week 8 was calculated as the daily mean of the daily frequencies during the week prior to the week 8 visit.
Time Frame: week 8 minus baseline
Measure: Mean (95% Confidence Interval); unit: Hot flashes/day
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 97 | 97
Hot flashes/day | -4.60 [-5.47 to -3.74] | -3.20 [-4.15 to -2.24]
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; Based on data from the Herbal Alternatives for Menopause (HALT) study, MsFLASH estimated that 90 women in each treatment group provide 90% power to detect a difference between drug and placebo with a 2-sided alpha of 0.025 to account for two primary outcomes of hot flash frequency and severity; Test type: Superiority or Other; p < 0.001, Regression, Linear — P values from comparison of Escitalopram vs placebo in a linear model of the outcome as a function of intervention group and adjusted for race, clinical center, baseline outcome, and visit (week 4 or week 8); Natural log transformations applied to hot flash frequencies for modeling assumptions

5. Primary Outcome: Daily Severity of Hot Flashes Assessed by Prospective Daily Diaries
Description: Daily hot flash severity scores were calculated by by selecting the highest severity rating for hot flashes or night sweats for each woman in each 24-hour day. The score was set to missing on on any day data were missing or or hot flashes equaled 0. The daily mean of daily ratings for the first 2 screening weeks is reported.
  Hot flash severity was rated as 1 (mild), 2 (moderate), or 3 (severe) as adopted from the Study of Women Across the Nation (SWAN).
Time Frame: Baseline
Population: Hot flash severity was rated as 1 (mild), 2 (moderate), or 3 (severe) as adapted from the Study of Women Across the Nation (SWAN).
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 104 | 101
Scores on a scale | 2.16 [2.07 to 2.24] | 2.19 [2.10 to 2.28]

6. Secondary Outcome: Change in Daily Hot Flash Bother Between Baseline and Week 4 as Recorded on Daily Diaries
Description: Change in daily hot flash bother was calculated as the mean difference between baseline and week 4. Baseline was calculated as the daily mean of the highest daily bother ratings during the first two screening weeks. Week 4 was calculated as the daily mean of the highest of the daily bother ratings during the week prior to the week 4 visit.
  Hot flash bother was rated as 1 (none), 2 (a little), 3 (moderately), or 4 (a lot) as adopted from the Study of Women Across the Nation (SWAN).
Time Frame: week 4 minus baseline
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 100 | 97
Scores on a scale | -0.59 [-0.73 to -0.45] | -0.29 [-0.41 to -0.16]

7. Primary Outcome: Change in Daily Severity of Hot Flashes Between Baseline and Week 4 as Assessed by Prospective Daily Diaries
Description: Change in daily hot flash severity from baseline to week 4 was calculated as the mean difference in hot flash severity ratings between baseline and week 4. Baseline was calculated as the daily mean from the first two weeks of hot flash severity ratings. Week 4 severity ratings were calculated as the daily mean from the ratings for the week prior to the week 4 visit.
  Hot flash severity was rated as 1 (mild), 2 (moderate), or 3 (severe) as adopted from the Study of Women Across the Nation (SWAN).
Time Frame: week 4 minus baseline
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 100 | 97
Scores on a scale | -0.43 [-0.54 to -0.33] | -0.23 [-0.34 to -0.13]

8. Primary Outcome: Change in Daily Severity of Hot Flashes Between Baseline and Week 8 as Assessed by Prospective Daily Diaries
Description: Change in daily hot flash severity between baseline & week 8 was calculated as mean difference. Baseline severity ratings were calculated as daily mean ratings for the first two screening weeks pre-baseline. Week 8 severity ratings were calculated as daily mean ratings during the week before week 8. Modified intention to treat analysis included all randomized participants who provided diary data, which were analyzed regardless of adherence to treatment assignment. Hot flash severity was rated as 1 (mild), 2 (moderate), or 3 (severe) as adopted from the Study of Women Across the Nation (SWAN).
Time Frame: week 8 minus baseline
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 96 | 96
Scores on a scale | -0.53 [-0.64 to -0.40] | -0.30 [-0.42 to -0.17]
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Linear — [p-value comment as in outcome 4, analysis 1]; Natural log transformations applied to hot flash frequencies for modeling assumptions

9. Secondary Outcome: Secondary Outcome: Change in Daily Hot Flash Bother Between Baseline and Week 8 as Recorded on Daily Diaries
Description: Change in daily hot flash bother between baseline & week 8 was calculated as mean difference. Baseline daily bother was the mean of the highest daily ratings for two screening weeks pre-baseline. Week 8 bother was daily mean of the highest daily bother ratings during the week before week 8. Modified intention to treat analysis included all randomized participants who provided diary data, which were analyzed regardless of adherence to treatment assignment. Hot flash bother was rated as 1 (none), 2 (a little), 3 (moderately), 4 (a lot) as adopted from the Study of Women Across the Nation (SWAN).
Time Frame: week 8 minus baseline
Population: Twice daily rating for bother using response categories from the Study of Women Across the Nation (SWAN): 1 (not at all), 2 (very little), 3 (moderately), 4 (a lot).
  Modified intention to treat analysis included all randomized participants who provided diary data, which were analyzed regardless of adherence to treatment assignment.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 96 | 96
Scores on a scale | -0.63 [-0.78 to -0.49] | -0.39 [-0.55 to -0.24]
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Linear

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 8 week treatment period.
Description: Participants were assessed at baseline for symptoms using a a self-administered questionnaire listing 12 common selective serotonin reuptake inhibitor (SSRI) adverse events. Newly emergent adverse events were collected at each study visit (week 4, week 8) using a self-administered questionnaire listing 12 common SSRI adverse events.
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/101
Other Adverse Events (participants affected / at risk) | 54/104 | 62/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=104) | Placebo (N=101)
Fatigue, tiredness (General disorders) | 14 (14) | 14 (14)
Difficulty sleeping/insomnia (General disorders) | 9 (9) | 10 (10)
Drowsiness (General disorders) | 14 (14) | 13 (13)
Increased sweating (General disorders) | 7 (7) | 9 (9)
Dry mouth (General disorders) | 11 (11) | 12 (12)
Stomach or intestinal problems (General disorders) | 10 (10) | 18 (18)
Nausea or vomiting (General disorders) | 11 (11) | 5 (5)
Decreased sexual desire/ability (General disorders) | 7 (7) | 8 (8)
Headache (General disorders) | 8 (8) | 11 (11)
Vivid dreams (General disorders) | 8 (8) | 9 (9)
Appetite changes (General disorders) | 6 (6) | 4 (4)
Other symptoms (General disorders) | 4 (4) | 10 (10)
Dizziness/lightheadedness (General disorders) | 3 (3) | 7 (7)

LIMITATIONS AND CAVEATS:
Although this was a community-based sample, the volunteers may be a select group motivated to seek treatment. An 8-week trial is brief, but data indicate that this interval is sufficient to determine long-term efficacy of a nonhormonal compound.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No